CLINICAL TRIAL: NCT00507767
Title: A Phase 2 Study of Dasatinib in Head and Neck Squamous Cell Carcinoma
Brief Title: Dasatinib in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00227; NCI-2009-00227 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000559148; 2006-0571 (Other: M D Anderson Cancer Center); 7815 (Other: CTEP); N01CM62202 (NIH); P30CA016672 (NIH); NCT00513227 (obsolete NCT alias)
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Dasatinib

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO or via PEG tube BID. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib; Procedure: pharmacological study; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: dasatinib — Given PO or via PEG tube
  Other Names: BMS-354825; Sprycel
Procedure: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well dasatinib works in treating patients with head and neck cancer that has come back or spread to other areas of the body. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 12-week progression-free survival rate and the objective response rate, as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, in patients with recurrent or metastatic squamous cell carcinoma of the head and neck treated with dasatinib.

SECONDARY OBJECTIVES:

I. To define metabolic response rate by positron emission tomography (PET) scan at 0, 8, and 12 weeks.

II. To define overall survival distribution from initiation of dasatinib. III. To define duration of response. IV. To determine if there is a correlation between clinical benefit from dasatinib (defined as disease response or stabilization) and pharmacokinetics, pharmacodynamics (phosphorylated Src [pSrc] expression in platelets), or changes in serum levels of cytokines, growth factors, and growth factor receptors relevant to the Src signaling pathway.

V. To examine the relationship between clinical benefit and mammary tumor and squamous cell carcinoma-associated protein (EMS1) gene amplification and cortactin expression levels in tumor tissue prior to therapy and the modulation of cortactin levels by treatment.

VI. To compare the effects of dasatinib on apoptosis by terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL) assay in tumor tissues comparing pre- and post-treatment biopsies.

VII. To assess the tolerability of dasatinib in this patient population. VIII. To describe the pharmacokinetic (PK) profile and relative bioavailability of dasatinib suspension in patients receiving the drug through percutaneous gastrostomy tube.

IX. To descriptively assess safety, toxicity, and efficacy of dasatinib crushed and administered by feeding tube.

OUTLINE:

Patients receive dasatinib orally (PO) or via percutaneous gastrostomy (PEG) tube twice daily (BID). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically proven squamous cell carcinoma of the head and neck that is recurrent after surgery and/or radiation therapy or chemoradiation therapy or is metastatic and disease must be measurable by RECIST criteria
* Patients must have measurable disease as defined by RECIST criteria
* Patients have received =< 1 prior chemotherapeutic regimen for recurrent or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin (Hgb) >= 9.0 g/dL
* Total bilirubin =< 1.5 X upper limit of normal
* Albumin >= 2.5 g/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 1.5 X upper limit of normal
* Creatinine =< 3 mg/dl
* Paraffin embedded tumor tissue that is appropriate for immunohistochemistry (IHC) and fluorescent in situ hybridization (FISH) analysis must be available or patient must be amenable to biopsy to obtain tissue for the study
* Ability to understand and the willingness to sign a written informed consent document
* Patient must not be pregnant or breastfeeding; all sexually active females of child-bearing potential and all sexually active males with sexual partners of child-bearing potential should practice contraception (e.g. barrier, hormonal, intrauterine device [IUD]) or sexual abstinence while in the study and for two months following completion of therapy
* Brain metastases permitted provided the patient does not require anticonvulsants or corticosteroids, or has been off them at least 7 days; patients with brain metastases must be either > 4 weeks beyond cranial irradiation or must be felt not to require it at that time
* The patient's O2 saturation must be >= 92% on room air

Exclusion Criteria:

* Chemotherapy or palliative radiotherapy for recurrent and/or metastatic disease within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or failure to recover to at least grade 1 from adverse events due to agents administered more than 4 weeks earlier; concomitant chemoradiation therapy within 6 weeks prior to entering the study or failure to recover to at least grade 1 from adverse events due to agents administered more than 4 weeks earlier
* Other anti-neoplastic agents, i.e., cytotoxic chemotherapy, immunotherapy, radiotherapy or investigational therapy, used to treat the primary disease will not be allowed during the study; local radiation (excluding radiotherapy to the target lesion) for supportive reasons involving a small radiation field may be allowed
* Patient has a history of uncontrolled or severe medical disease which could compromise participation in the study such as uncontrolled diabetes (fasting blood glucose > 200 mg/dl), uncontrolled hypertension (systolic blood pressure [BP] > 160 or diastolic BP > 100 mmHg), severe infection (bacterial infection requiring intravenous [IV] antibiotics or human immunodeficiency virus [HIV]), angina at rest, congestive heart failure New York Heart Association (NYHA) class III or IV, ventricular arrhythmias requiring therapy, myocardial infarction within 6 months, > grade 2 neuropathy
* Patients may not be receiving any other investigational agents
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; efforts should be made to switch patients with gliomas or brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications
* Echocardiogram less than institutional normal measured by echocardiogram for subjects with history of congestive heart failure, symptoms of congestive heart failure, clinical evidence suggesting impaired cardiac function
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged correct QT interval (QTc) > 480 msec (Fridericia correction)
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* Pregnant women and women who are currently breast-feeding may not participate in this study; all women of childbearing potential must have a negative pregnancy test within 72 hours prior to enrolling in the study; postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patients having pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 24, 2007 to February 26, 2009. Al recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Dasatinib: 100 mg orally twice daily
Period: Overall Study
Arm/Group | Dasatinib
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 54 (10) [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival at 12-weeks
Description: Progression-free survival (PFS) is defined as stable disease or better. Participants who have received at least one dose of dasatinib and who die or leave the study before 12 weeks will be counted as having progressive disease.
Time Frame: At 12-weeks
Population: Analysis per protocol.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 15
participants | 1 [.2 to .05]

ADVERSE EVENTS:
Time Frame: Treatment period three 4-week cycles for total of 12 weeks with follow up every 2 cycles following first cycle. Study data collection period for all participants was 18 months.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=15)
Dehydration (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Toxicity (General disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=15)
Anorexia (General disorders) | 2
nausea/vomiting (Gastrointestinal disorders) | 15
diarrhea (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
dehydration (General disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
edema: limb (General disorders) | 3
Hearing (without monitoring) (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 1 — With normal Absolute neutrophil count (ANC)
Pain (bone) (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less